CLINICAL TRIAL: NCT03239912
Title: The Effects of Combined Treatment With Low-level Laser and Functional Appliances on the Correction of Class II Malocclusion: A Randomized Controlled Trial
Brief Title: Treatment of Class II Malocclusion Combined With Low-level Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-05-2017
Record Dates: First submitted 2017-07-28; First posted 2017-08-04 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion, Angle Class II
Keywords: Low-level laser; functional treatment; twin-block; RCT
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin-block group (Experimental): Functional treatment will be applied using the Twin-block appliance.
  Interventions: Device: Twin-block appliance
- Twin-block combined with low level laser (Experimental): Functional treatment will be applied using the Twin-block appliance combined with low level laser.
  Interventions: Device: Twin-block appliance; Other: Low level laser

INTERVENTIONS:
Device: Twin-block appliance — Functional treatment will be achieved using the Twin-block appliance
Other: Low level laser — Functional treatment will be combined with low-level laser therapy on the TMG region
  Arms: Twin-block combined with low level laser

SUMMARY:
This experimental study will evaluate the effect of combined treatment with low-level laser and functional appliances (twin-block) on the correction of Class II malocclusion, compared with the control group treated with functional appliances (twin-block) only.

The study sample will consist of 40 patients with Class II malocclusion. The sample will be allocated randomly into two groups: a control group and an experimental group.

Functional appliance (twin-block) will be applied for all patients. Low-level laser will be applied for the experimental group only. The skeleto-dental changes occurring after functional treatment will be assessed using cephalometric radiographs; pre- and post- treatment changes for each group will be evaluated individually.

DETAILED DESCRIPTION:
Class II malocclusion is considered as the most common malocclusion between patients.

Recently low-level laser enters the world of dentistry, some studies assessed the effect of low-level laser on the growth of mandibles and condyles in animals and showed that there is a good effect of laser on the mandible growth.

This study will evaluate the effect of low-level laser on the growth of the mandible and the duration of functional treatment.

Twin-block will be applied in two groups: The control group will receive the twin-block only, and the experimental group will receive the twin-block combined with low-level laser therapy on the TMG region.

Cephalometric radiographs will be gotten before and after functional treatment to evaluate the dento-skeletal changes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class II malocclusion because of mandibular retrognathia
* ANB > 4
* Overjet > 5
* SNB < 78

Exclusion Criteria:

* Poor oral hygiene
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Reason of contraindication of functional treatment

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
The duration of functional treatment | After functional treatment which will take approximately 8 months
  The duration of the functional treatment will be measured and compared between groups.

SECONDARY OUTCOMES:
Dentoskeletal effects of the functional treatment | Changes will be evaluated before and after functional treatment which will take approximately 8 months
  Dentoskeletal changes before and after functional treatment combined with Low-level Laser compared with those of the control group (SNA, SNB, ANB, Overjet ,…etc) using lateral cephalometric radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Abtahi M, Poosti M, Saghravanian N, Sadeghi K, Shafaee H. The effect of low level laser on condylar growth during mandibular advancement in rabbits. Head Face Med. 2012 Feb 23;8:4. doi: 10.1186/1746-160X-8-4. PMID 22361310
- [Background] Angeletti P, Pereira MD, Gomes HC, Hino CT, Ferreira LM. Effect of low-level laser therapy (GaAlAs) on bone regeneration in midpalatal anterior suture after surgically assisted rapid maxillary expansion. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Mar;109(3):e38-46. doi: 10.1016/j.tripleo.2009.10.043. PMID 20219584
- [Background] Oksayan R, Sokucu O, Ucuncu N. The effects of low-level laser therapy on condylar growth with a mandibular advancement appliance in rats. Photomed Laser Surg. 2015 May;33(5):252-7. doi: 10.1089/pho.2014.3870. Epub 2015 Apr 13. PMID 25867096
- [Background] Seifi M, Maghzi A, Gutknecht N, Mir M, Asna-Ashari M. The effect of 904 nm low level laser on condylar growth in rats. Lasers Med Sci. 2010 Jan;25(1):61-5. doi: 10.1007/s10103-009-0651-x. Epub 2009 Feb 24. PMID 19238504